CLINICAL TRIAL: NCT04696354
Title: Intravascular Ultrasound-Guided Intervention for Venous Leg Ulcers
Brief Title: Intravascular Ultrasound-Guided Intervention for Venous Leg Ulcers (IGuideU)
Acronym: IGuideU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped due to ongoing enrollment challenges.
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IGT_IGD_VLU_2020_10876; 200202 (Other: IGTD Protocol no.)
Record Dates: First submitted 2020-12-14; First posted 2021-01-06 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2023-01

CONDITIONS: Venous Ulcer of Leg
Keywords: VLU; venous leg ulcer; ulcer; venous leg wound; venous stenting; IVUS; DVO
MeSH Terms: conditions — Varicose Ulcer; Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Interrogation Arm (Other): patients will first be evaluated with MPV (limited to 3 views). The prescribed course of treatment based on the MPV results will be documented and patients will then be evaluated using IVUS. A treatment plan based on IVUS results will be compared with the MPV guided treatment plan and any differences will be documented. Any patients determined to still require venous stenting based on IVUS results will be stented accordingly using IVUS to guide stent placement.
  Interventions: Diagnostic Test: IVUS
- Deferred Interrogation Arm (Other): Deferred Interrogation Guidelines for this study are as follows:
  Mandate:
  • Continued compression therapy/stockings as prescribed.
  Allow:
  * Periodic leg elevation.
  * Sclerotherapy under ulcer bed.
  * Recommend mechanical debridement as needed.
  * Wound biopsy if evidence of infection.
  * Systemic antibiotics if patient is diagnosed with an infection, avoid prophylactic prescription.
  * Pain management medication (Pentoxifylline/Trental) allowed but not recommended
  * Topical antimicrobial as needed.
  Prohibit:
  * Negative pressure systems.
  * Artificial and/or autologous skin grafting within first 3 months after randomization and within the first 3 months for subjects that crossover from deferred interrogation to the interrogation arm.
  Interventions: Other: Continued Compression Therapy/Stockings

INTERVENTIONS:
Diagnostic Test: IVUS — Those who are randomized to the interrogation arm will have diagnostic imaging performed by IVUS to determine their treatment plan.
  Arms: Interrogation Arm
Other: Continued Compression Therapy/Stockings — Those who are randomized to the deferred interrogation arm while continue compression therapy as prescribed.
  Arms: Deferred Interrogation Arm

SUMMARY:
This clinical study is a global, prospective, multi-center, randomized controlled trial to determine if the use of intravascular ultrasound (IVUS) as an adjunctive imaging modality and as an interventional treatment guide will result in a more accurate diagnosis of deep vein occlusion (DVO), will guide optimal therapy, and will provide better clinical outcomes with reduced cost of care for patients presenting with persistent venous leg ulcers (VLUs).

DETAILED DESCRIPTION:
This study will be conducted in 266 subjects presenting with venous ulcers that have previously undergone treatment for superficial of and/or perforator venous disease, if clinically indicated, followed by at least 3 months of prescribed compression therapy prior to screening.

There are 6 study visits for each subject that will be completed over a period lasting approximately 24 months. Subjects will undergo a baseline/screening assessment (visit 1) followed by an interrogation procedure (visit 2) if the subject is enrolled into the interrogation arm. If the subject is randomized to the deferred interrogation arm, he/she will have a hospital/office visit in lieu of the interrogation procedure, which will be considered visit 2. For statistical purposes, the wound assessment performed at the index procedure/hospital visit will be considered the baseline measurement. 30±14 days and 90±14 days after Visit 2, the subject will return to the office for a 1- and 3-month follow-up visit, respectively. The subjects will return at 6- and 12-months post-index procedure/Visit 2 for follow-up assessments. The follow-up period for this study will be approximately 24 months, with a phone call only at 24-months post-index procedure/visit 2.

The clinical study has a planned enrollment period of 36 months and a planned study duration period of 5.17 years

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 85 years of age.
* Able and willing to participate and comply with the protocol, including the defined follow-up schedule, by signing an Institutional Review Board (IRB) or Ethics Committee approved informed consent form.
* Active venous leg ulcer (CEAP C6).
* Previously completed treatment for clinically significant reflux in the superficial and/or perforator venous system of the target limb at least 3 months prior to enrollment, if clinically indicated.
* Completed at least 3 months of prescribed compression therapy after any ablation.
* Palpable dorsalis pedis or posterior tibial artery (DP/PT) pulses at ipsilateral foot or ankle brachial index (ABI) ≥0.8.
* Be able to ambulate unassisted or with non-motorized assistive devices.
* Current VLU present ≤48 months.

Exclusion Criteria:

* Patient is known pregnant or breast-feeding or planning to become pregnant in the following year.
* If antiplatelet and anticoagulation therapy cannot be tolerated.
* Previous venous stent implantation involving the target limb, target lesion, or inferior vena cava.
* Previous venovenous bypass surgery involving the target limb.
* Previous endovascular recanalization of the target lesion segment.
* Known metal allergy precluding stent implantation.
* Known or suspected to have inadequate inflow to support stent patency in the target limb.
* Active cancer diagnosis.
* Known positive test for COVID-19 (Sars-CoV-2) within the last 2 weeks and actively symptomatic.
* Known or suspected venous outflow obstruction caused by tumor compression/encasement with or without thrombus.
* Known allergy to contrast media that cannot adequately be pre-medicated prior to study procedure.
* Known renal dysfunction (defined as eGFR <30mL/min/1.73m2) that would preclude adequate contrast usage.
* Diagnosed with right heart failure/pulmonary hypertension.
* Has known clinically significant abnormal platelet count outside laboratory reference ranges.
* Has known clinically significant abnormal white blood cell count (WBC), fever, sepsis or positive blood culture.
* Organ transplant requiring immunosuppressant therapy.
* Unstable angina pectoris, or myocardial infarction within 30 days and/or hemorrhagic stroke within 3 months.
* Subjects with an active diagnosis of osteomyelitis of the ipsilateral limb.
* Previous or planned surgical or catheter-based procedure on index leg within 30 days before or 30 days after the index procedure.
* Active participation in another investigational drug or device study.
* Subject has any condition, which, in the opinion of the investigator, precludes the subject from participation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Black, MD, Principal Investigator — St. Thomas and Guys Hospital; Paul Gagne, MD, Principal Investigator — Vascular Care CT, PLLC
Locations (17):
- United States (8):
  - Vascular Care Connecticut, Darien, Connecticut
  - Florida Cardiology, P.A., Winter Park, Florida
  - Northwestern, Chicago, Illinois
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Vein Center of Southwest Louisiana, Lake Charles, Louisiana
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - NYU Langone Health, New York, New York
  - Atrium Health, Charlotte, North Carolina
- Australia (2):
  - Wollongong Hospital, Wollongong, New South Wales
  - Royal Perth Hospital, Perth, Western Australia
- France (3):
  - CHU Strasbourg, Strasbourg, Alsace
  - CH Vichy, Vichy, Bourbonnais
  - C.H.U. Dijon, Dijon
- Klinikum Hochsauerland GmbH, Arnsberg, North Rhine-Westphalia, Germany
- United Kingdom (3):
  - Northwick Park Hospital, Harrow, London
  - Royal Free London NHS Foundation Trust, Hampstead
  - Guys and St. Thomas' Hospital, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No analysis performed. Study was terminated due to slow enrollment. Only 12 enrollments of the required 266 subjects.
Pre-assignment Details: For the small number of enrolled patients no data was collected for analysis. No outcome measures to report.
Groups:
- Deferred Interrogation Arm: Deferred Interrogation Guidelines for this study are as follows:
  Mandate:
  • Continued compression therapy/stockings as prescribed.
  Allow:
  * Periodic leg elevation.
  * Sclerotherapy under ulcer bed.
  * Recommend mechanical debridement as needed.
  * Wound biopsy if evidence of infection.
  * Systemic antibiotics if patient is diagnosed with an infection, avoid prophylactic prescription.
  * Pain management medication (Pentoxifylline/Trental) allowed but not recommended
  * Topical antimicrobial as needed.
  Prohibit:
  * Negative pressure systems.
  * Artificial and/or autologous skin grafting within first 3 months after randomization and within the first 3 months for subjects that crossover from deferred interrogation to the interrogation arm.
  Continued Compression Therapy/Stockings: Those who are randomized to the deferred interrogation arm while continue compression therapy as prescribed.
Period: Overall Study
Arm/Group | Interrogation Arm | Deferred Interrogation Arm
Started | 6 | 6
Completed | 0 | 0
Not Completed | 6 | 6
Not completed — Study termination | 6 | 6

BASELINE CHARACTERISTICS:
Population: No data collected for analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Interrogation Arm | Deferred Interrogation Arm | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Full Range); unit: years] — Population: No statistical analysis was performed.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: No statistical analysis was performed.
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: No statistical analysis was performed
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3
  United Kingdom | 4 | 4 | 8
  France | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate of Detection and Difference in Complete Ulcer Healing Between the Interrogation Group and the Deferred Interrogation Group
Description: Rate of detection and difference in complete ulcer healing between the interrogation group and the deferred interrogation group at 3 months. Complete ulcer healing is defined by 100% epithelialization of the venous ulcer. Healing will not be assumed for any area of the wound where a scab is present.
Time Frame: 3 months
Population: No data was collected for analysis. No outcome data to report.
Groups:
- Deferred Interrogation: Deferred Interrogation Guidelines for this study are as follows:
  Mandate:
  • Continued compression therapy/stockings as prescribed.
  Allow:
  Periodic leg elevation. Sclerotherapy under ulcer bed. Recommend mechanical debridement as needed. Wound biopsy if evidence of infection. Systemic antibiotics if patient is diagnosed with an infection, avoid prophylactic prescription.
  Pain management medication (Pentoxifylline/Trental) allowed but not recommended Topical antimicrobial as needed.
  Prohibit:
  Negative pressure systems. Artificial and/or autologous skin grafting within first 3 months after randomization and within the first 3 months for subjects that crossover from deferred interrogation to the interrogation arm.
Arm/Group | Interrogation Arm | Deferred Interrogation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: This study was terminated due to slow enrollment, only 12 of 266 subjects were enrolled. No data was collected for statistical analysis.
Description: This study was terminated due to slow enrollment, only 12 of 266 subjects were enrolled. No data was collected for statistical analysis.
Arm/Group | Interrogation Arm | Deferred Interrogation Arm
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This study was terminated due to slow enrollment, only 12 of 266 subjects have been enrolled. Because enrollment in this clinical trial did not reach the target number of subjects needed to achieve target power, no data was collected. No statistical analysis information will be submitted for the outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT04696354/Prot_SAP_000.pdf